CLINICAL TRIAL: NCT02978339
Title: An Open-Label Pilot Study Evaluating the Safety and Efficacy of Curcumin in Patients With Primary Sclerosing Cholangitis
Brief Title: A Study Evaluating the Safety and Efficacy of Curcumin in Patients With Primary Sclerosing Cholangitis (PSC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John E. Eaton (Other)
Collaborators: EuroPharma, Inc. (Industry)
Responsible Party: Sponsor-Investigator, John E. Eaton, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-002660
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Curcumin (Experimental): Subjects will receive one 750 mg softgel by mouth twice a day for 12 weeks. Each each 750 mg CuraMed® softgel supplies 500 mg of highly bioavailable BCM-95 curcumin.
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — Subjects will receive one 750 mg softgel by mouth twice a day for 12 weeks. Each each 750 mg CuraMed® softgel supplies 500 mg of highly bioavailable BCM-95 curcumin.
  Other Names: CuraMed® softgel

SUMMARY:
The purpose of this study is to determine whether curcumin, a drug and naturally-occurring plant compound, is safe and effective in the treatment of primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary sclerosing cholangitis (PSC) established by all of the following criteria:

  * Alkaline phosphatase >1.5x upper limit of normal for at least 6 months prior to study enrollment
  * Cholangiography demonstrating intrahepatic and/or extrahepatic biliary dilation, beading, and/or strictures consistent with PSC
  * Liver histology (if available for review) consistent with or diagnostic of PSC
* Women of child-bearing potential willing to use birth control for the duration of the study.

Exclusion Criteria:

* Treatment with any investigational agents within three months prior to or during the study
* Treatment with systemic antibiotics, azulfidine, systemic corticosteroids, colchicine, methotrexate, azathioprine, cyclosporine, chlorambucil, budesonide, pentoxifylline, tacrolimus, or vitamin E within three months prior to or during the study.
* Concomitant treatment with NSAIDS, antiplatelet agents, antihyperlipidemics, and anticoagulant warfarin.
* Anticipated need for liver transplant within one year as determined by Mayo PSC risk score (<80% one-year survival without transplant)
* Active drug or alcohol use
* Findings suggestive of liver disease of an alternative or concomitant etiology, such as chronic alcoholic liver disease, chronic hepatitis B or C infection, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or secondary sclerosing cholangitis (e.g., post-liver transplantation biliary stricture)
* Pregnancy or lactation
* Any condition that, in the opinion of the investigator, would interfere with the patient's ability to complete the study safely or successfully.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas F LaRusso, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Curcumin
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Curcumin
Number analyzed (Participants) | 15
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 46 [39 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15
Primary Sclerosing Cholangitis Duration [Mean (Inter-Quartile Range); unit: years] | 9.00 [4 to 13]
Inflammatory Bowel Disease Present [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Alkaline Phosphatase (SAP)
Description: Number of subjects who experience a reduction of Serum Alkaline Phosphatase (SAP) to less than 1.5 x Upper Limit of Normal or a 40% reduction between baseline and week 12.
Time Frame: baseline, 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Curcumin
Number analyzed (Participants) | 15
Participants | 3
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = .03, t-test, 2 sided

2. Secondary Outcome: Change in Serum Aspartate Aminotransferase (AST)
Description: AST is an enzyme found in high amounts in liver, heart, and muscle cells. This test is mainly done along with other tests such as alkaline phosphatase and bilirubin to diagnose and monitor liver disease. This test evaluates hepatocyte integrity, as serum levels of this enzyme rise in response to a variety of forms of injury to hepatic cells. The normal range is 10 to 40 Unit/Liter (U/L)
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Curcumin
Number analyzed (Participants) | 15
U/L | 78 [48 to 119]
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = 0.59, t-test, 2 sided

3. Secondary Outcome: Change in Total Bilirubin
Description: Bilirubin is a yellowish pigment found in bile, a fluid made by the liver. A small amount of older red blood cells are replaced by new blood cells every day. Bilirubin is left after these older blood cells are removed. The liver helps break down bilirubin so that it can be removed from the body in the stool. The normal range for total bilirubin is 0.3 to 1.9 milligrams/deciliter (mg/dL)
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Curcumin
Number analyzed (Participants) | 15
mg/dL | 0.6 [0.5 to 1.4]
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = 0.91, t-test, 2 sided

4. Secondary Outcome: Change in C-Reactive Protein (CRP)
Description: C-reactive protein is a substance produced by the liver in response to inflammation. Normal CRP levels are below 3.0 milligrams/Liter (mg/L)
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Curcumin
Number analyzed (Participants) | 15
mg/L | 3.4 [1.5 to 9.1]
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = 0.41, t-test, 2 sided

5. Secondary Outcome: Change in Mayo Primary Sclerosing Cholangitis (PSC) Risk Score
Description: The Mayo Risk Score (R) = (0.0295 * (age in years)) + (0.5373 * natural logarithm(total bilirubin in mg/dL)) - (0.8389 * (serum albumin in g/dL)) + (0.5380 * natural logarithm(AST in IU/L) + (1.2426 * (points for variceal bleeding)) where:
  AST = serum aspartate aminotransferase level, Points for variceal bleeding: 0 if none, 1 if present. Each unit increase in the Mayo Risk Score (R) is associated with a 2.5-fold increase in the risk of death. Most references to the score round the coefficients to 2 decimal places. The score shows very slight upward slope over time in stable patients, but during the terminal phase it shows an acceleration in progression.
Time Frame: Baseline, 12 weeks
Population: Twelve subjects completed questionnaires. Three subjects did not complete questionnaires
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Curcumin
Number analyzed (Participants) | 12
score on a scale | 0.54 [-0.17 to 0.63]
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = .15, t-test, 2 sided

6. Secondary Outcome: Change in Fatigue Severity
Description: Fatigue will be measured by a Modified Fatigue Impact Scale (MFIS). This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items. Subjects rate on a 5-point scale with 0 = never to 4 = almost always. The total score for the MFIS is the sum of the scores for the 21 items ranging from score of 0-84. Higher numbers indicate greater fatigue.
Time Frame: Baseline, 12 weeks
Population: Twelve subjects completed questionnaires. Three subjects did not complete questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Curcumin
Number analyzed (Participants) | 12
score on a scale | 8.00 [4.00 to 23.00]
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = .06, t-test, 2 sided

7. Secondary Outcome: Change in Pruritus
Description: Pruritus will be measured by the 5-D itch Scale. The 5-D itch scale was developed as a brief but multidimensional questionnaire designed to be useful as an outcome measure in clinical trials." The five dimensions are degree, duration, direction, disability and distribution. The duration, degree and direction domains each include one item, while the disability domain has four items. All items of the first four domains were measured on a five-point Likert scale (1 = Not present/resolved/never, 5 = Unbearable/getting worse/always).The distribution domain included 16 potential locations of itch, including 15 body part items and one point of contact with clothing or bandages.The scores of each of the five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritus) and 25 (most severe pruritus)
Time Frame: Baseline, 12 weeks
Population: Twelve of the subjects completed questionnaires. Three subjects did not complete questionnaires
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Curcumin
Number analyzed (Participants) | 12
score on a scale | 8.00 [7.50 to 14.50]
Statistical Analysis 1: Comparison: Curcumin; Test type: Superiority; p = .93, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 12 weeks
Arm/Group | Curcumin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curcumin (N=15)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Blood Bilirubin increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT02978339/Prot_SAP_000.pdf